CLINICAL TRIAL: NCT01264783
Title: Phase I, Double-blind, Randomized, Placebo-controlled, Single-center Study to Assess the Safety and Tolerability of RNS60 Administered Intravenously to Healthy Subjects
Brief Title: Safety and Tolerability of RNS60 Given by IV to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11.1.1.H1
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-09

CONDITIONS: Myocardial Infarct
MeSH Terms: conditions — Myocardial Infarction | interventions — RNS60

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RNS60 (Experimental): RNS60
  Interventions: Drug: RNS60
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RNS60 — RNS60 for intravenous administration
  Arms: RNS60
Drug: Placebo — 0.9% normal saline for injection
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of RNS60 administered intravenously to healthy subjects. 12 subjects will receive RNS60 or placebo at three escalating rates for 48 hours for each rate.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18-55 years
* Minimum body weight of 60 kg
* BMI of 18-32 kg/m2
* Able to execute informed written consent

Exclusion Criteria:

* A chronic or acute disease that might interfere with the evaluation of the safety of RNS60
* Current or prior malignancies (excluding history of treated non-melanoma skin carcinoma)
* Positive viral serology test for HBsAG, Hep C antibody, Hep A IgM, or HIV
* Use of any prescription medications within 2 weeks of the first day of dosing
* Significant organ dysfunction, including cardiac, renal, liver, CNS, pulmonary, vascular, GI, endocrine or metabolic
* Treatment with monoclonal antibody therapy within 5 half-lives prior to the first dose of study medication
* Treatment with any investigational drugs or therapies within 30 days (or 5 half-lives, whichever is greater) prior to the first dose of study medication
* Abnormal pre-admission vital signs, physical exam, clinical laboratory, or any safety variable considered clinically significant for this population by the PI
* Subject is considering or has scheduled any surgical procedure during participation in study
* History of alcohol and/or dug abuse within 1 year prior to first dose of study medication
* Subject has donated plasma or blood within 30 days prior to first dose of study medication
* Subject requires treatment with any medications, either prescription or nonprescription, including dietary supplements or herbal medications, within 14 days prior to the first dose of study medication. Exceptions are nonprescription topical medications (that are not systemically absorbed), acetaminophen, or vitamins at recommended daily doses (not mega dose vitamins)
* A positive qualitative urine drug or alcohol test
* Concurrent enrollment in any other clinical trial
* Subject is judged by PI or Medical Monitor to be inappropriate for the study -
* Subject has Gilbert's syndrome
* Subject has estimated creatinine clearance at screening of <90 mL/min.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Tolerability | 6 days
  Safety and tolerability of RNS60 administered by IV infusion to healthy volunteers.

SECONDARY OUTCOMES:
Biomarkers | 6 days
  Analysis of blood samples for various biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Craven, M.D., Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles, Inc., Overland Park, Kansas, United States